CLINICAL TRIAL: NCT05061680
Title: Endoscopic Papillary Short Duration Large Balloon Dilatation for Removal of Large Bile Duct Stones: a Prospective Multicenter Study of Short and Long-term Adverse Events
Brief Title: Quick Large Balloon Dilatation for Removal of Large Bile Duct Stones (SHODBADI)
Acronym: SHODBADI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Mia Rainio, Principal Investigator, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Largeballoon dilation
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Pancreatitis, Acute; Bleeding; Cholangitis
MeSH Terms: conditions — Pancreatitis; Hemorrhage; Cholangitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- short sphincterotomy +Short duration papillary large balloon dilation (Active Comparator): Patients with short sphincterotomy
  Interventions: Device: endoscopic short duration papillary large balloon dilation
- full sphincterotomy + short duration papillary balloon dilation (Active Comparator): Patients with full lenght sphincterotomy
  Interventions: Device: endoscopic short duration papillary large balloon dilation
- previous sphincterotomy + short duration papillary balloon dilation (Active Comparator): Patients with previous sphincterotomy
  Interventions: Device: endoscopic short duration papillary large balloon dilation

INTERVENTIONS:
Device: endoscopic short duration papillary large balloon dilation — During the large balloon papillary dilation investigators follow the cholangiogram and stop the dilatation as soon as the disappearance of the waist of the papilla is noticed.

SUMMARY:
ESGE guidelines suggests 30-60 seconds endoscopic large balloon papillary dilation from the disappearance of the waist of the papilla.

The investigators have good results in stone removal with much quicker dilatations when the cholangiogram is followed and the dilation is finished as soon as the disappearance of the waist of the papilla is seen. This Scandinavian multicenter prospective study is especially interested in stone clearance rate and short and long-term adverse events such as pancreatitis, cholangitis, bleeding, perforations, residual biliary stones, and newly developing biliary stones.

DETAILED DESCRIPTION:
This study is planned as a multicenter Scandinavian prospective study including all the patients >18 years with >10mm diameter common bile duct stones visible in cholangiogram. Before ERCP all patient will be informed about this trial, and if they agree to participate this study, they need to give a written informed consent. The endoscopists will decide whether the first step will be large EST and stone extraction or small EST and dilatation. If simple EST does not success, the dilatation will remain as a rescue method. The diameter of dilatation balloon cannot exceed the diameter of common bile duct above the papilla. Cholangiogram is followed when papilla is dilated and the dilatation will be ended when the waist of the papilla disappears. The duration of the dilatation measured, but it does not define the ending of dilatation. All adverse events will be recorded one month and a year after the procedure.

Classification of the patients:

1. EST and stone extraction
2. EPLBD when EST and stone extraction did not succeed
3. Short EST and EPLBD

The investigators will collect the information of adverse events such as bleeding, pancreatitis, cholangitis with patient questionnaire as well as from the patient records one month and a year after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Common bile duct stone >10mm diameter

Exclusion Criteria:

* Altered anatomy after surgery (B II, Roux-en-Y reconstruction)
* Common bile duct cysts
* Acute pancreatitis
* Distal common bile duct stricture or tumor
* Coagulation disorders
* Ongoing coagulation medication
* Pregnancy
* Inability to give an informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of bleeding | 30 days
  need for additional intervention or need for blood transfusion and hemoglobin drop more than 2 gm/dL
Rate of pancreatitis | 30 days
  Plasma amylase rises >3 times the upper limit and newly developed stomach ace more than 24h
Rate of cholangitis | 30 days
  Fever >38

CONTACTS AND LOCATIONS:
Overall Officials: Mia Rainio, Md, PhD, Study Director — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No